CLINICAL TRIAL: NCT01401218
Title: Incidence, Risk Factors, and Risk Model of Acute Kidney Injury After Thoracic Aortic Surgery
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Sangmin M. Lee, Professor, Samsung Medical Center
Other Study IDs: 2011-06-077
Record Dates: First submitted 2011-07-21; First posted 2011-07-25 (Estimated); Last update posted 2013-12-25 (Estimated); Status verified 2013-12

CONDITIONS: Thoracic Aortic Surgery
Keywords: thoracic aortic surgery; acute kidney injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — Electronic Health Records

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- thoracic aortic surgery group: patients who underwent thoracic aortic surgery
  Interventions: Other: Electronic Medical Record (EMR) Review

INTERVENTIONS:
Other: Electronic Medical Record (EMR) Review — measurements of potential risk factors of acute kidney injury through the patients' previous medical record review.
  potential risk factors include previous history of hypertension, diabetes, cerebrovascular events, peripheral arterial disease, chronic obstructive pulmonary disease, recent myocardial infarction, coronary artery disease; preoperative glomerular filtration rate, preoperative creatinine level, preoperative cardiac ejection fraction reported on echocardiography, use of preoperative inotropics, use of deep hypothermic cardiac arrest, intraoperative colloid use, intraoperative blood product transfusion, total time of cardiopulmonary bypass,
  Other Names: Electronic Medical Record (EMR)

SUMMARY:
Postoperative acute kidney injury (AKI) is still one of the serious complications of thoracic aortic surgery, with incidence of 8 to 50 percent. Postoperative AKI significantly increases the morbidity and mortality of patients undergoing thoracic aortic surgery. Previous studies for AKI after DHCA reported confounding results due to different criteria of AKI. Therefore, the investigators tried to evaluate the incidence and risk factors of AKI after thoracic aortic surgery according to the diagnostic criteria and staging system of AKI reported from acute kidney injury network. The investigators also tried to develop a risk model with scoring system of AKI and evaluate the performance of the risk model.

DETAILED DESCRIPTION:
Significant improvement of morbidity and mortality has been achieved during last three decades since developing deep hypothermic circulatory arrest (DHCA). However,postoperative acute kidney injury (AKI) is still one of the serious complications of thoracic aortic surgery, with incidence of 8 to 50 percent. Postoperative AKI significantly increases the morbidity and mortality of patients undergoing thoracic aortic surgery. Previous studies for AKI after DHCA reported confounding results due to different criteria of AKI. Therefore, the investigators tried to evaluate the incidence and risk factors of AKI after thoracic aortic surgery according to the diagnostic criteria and staging system of AKI reported from acute kidney injury network (2007). The investigators also tried to develop a risk model with scoring system of AKI and evaluate the performance of the risk model.

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent thoracic aortic surgery during 1994 to 2010 period

Exclusion Criteria:

* patients who had previous renal failure before aortic surgery

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who underwent thoracic aortic surgery durung 1994 to 2010 period
Sampling Method: Non-Probability Sample
Enrollment: 799 (Actual)
Dates: Start 2011-07; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
presence of Acute kidney injury | 1 time, within 48 hours of aortic surgery
  diagnosis of AKI if the record of patient meet one of the below criteria
  1. abrupt (within 48 hours) reduction in kidney function currently defined as
  2. absolute increase in serum creatinine of more than or equal to 0.3 mg/dl (≥ 26.4 μmol/l),
  3. a percentage increase in serum creatinine of more than or equal to 50% (1.5-fold from baseline), or
  4. a reduction in urine output (documented oliguria of less than 0.5 ml/kg per hour for more than six hours)

CONTACTS AND LOCATIONS:
Overall Officials: Sangmin M. Lee, M.D.,Ph.D., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea